CLINICAL TRIAL: NCT07273474
Title: A Phase I, Open-label Trial in Two Parallel Parts to Investigate Mass Balance, Metabolism, and Basic Pharmacokinetics of BI 3000202 (C-14) Administered as Oral Solution (Part A) and to Investigate Absolute Bioavailability (BA) of BI 3000202 Administered as Film Coated Tablet Together With an Intravenous Microtracer Dose of BI 3000202 (C-14) (Part B) in Healthy Male and Female Participants
Brief Title: A Study in Healthy Men and Women to Test How BI 3000202 is Taken up and Processed by the Body
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1509-0010; 2023-510345-21-00 (Registry Identifier: CTIS); U1111-1301-4856 (Registry Identifier: WHO - International Clinical Trials Registry Platform (ICTRP))
Record Dates: First submitted 2025-11-27; First posted 2025-12-09 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part A (Experimental): Absorption, distribution, metabolism, and excretion (ADME)
  Interventions: Drug: BI 3000202; Drug: BI 3000202 [14C]-labelled
- Part B (Experimental): Bioavailability (BA)
  Interventions: Drug: BI 3000202; Drug: BI 3000202 [14C]-labelled

INTERVENTIONS:
Drug: BI 3000202 — BI 3000202 unlabelled
Drug: BI 3000202 [14C]-labelled — BI 3000202 [14C]-labelled

SUMMARY:
The purpose of this study is to find out how quickly and to what extent BI 3000202 is processed in the body.

The purpose of Part A is to find out how 3000202 moves through and exits the body of healthy people. The purpose of Part B is to find out how much BI 3000202 gets into the blood when participants take it as a tablet compared with when they get it as an infusion.

Adults between 18 and 55 years of age can take part if the study doctor determines they are healthy.

The doctors regularly check participants' health. To assess the study endpoints, the study staff takes blood, urine, and stool samples.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female of non-childbearing potential trial participants according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (blood pressure (BP), pulse rate (PR)), 12-lead electrocardiogram (ECG), and clinical laboratory tests
2. Age of 18 to 55 years (inclusive)
3. Body mass index (BMI) of 18.5 to 30 kg/m² (inclusive)
4. Signed and dated written informed consent in accordance with ICH-GCP and local legislation prior to admission to the trial

Exclusion Criteria:

1. Any finding in the medical examination (including BP, PR or ECG) deviating from normal and assessed as clinically relevant by the investigator
2. Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg (inclusive), diastolic blood pressure outside the range of 50 to 90 mmHg (inclusive), or pulse rate outside the range of 40 to 99 bpm (inclusive)
3. Any laboratory value outside the reference range that the investigator considers to be of clinical significance
4. Any evidence of a concomitant disease assessed as clinically significant by the investigator Further exclusion criteria apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2025-12-30 (Actual); Primary Completion 2026-03-05 (Estimated); Study Completion 2026-03-05 (Estimated)

PRIMARY OUTCOMES:
Part A: fe-urine, 0-tz (fraction excreted in urine as percentage of the administered dose over the time interval from 0 to the last quantifiable time point) | up to 21 days
Part A: fe-faeces, 0-tz (fraction excreted in faeces as percentage of the administered dose over the time interval from 0 to the last quantifiable time point) | up to 21 days
Part B: AUC0-∞ (area under the concentration-time curve of the analyte over the time interval from 0 extrapolated to infinity) | up to 6 days

SECONDARY OUTCOMES:
Part A: Cmax (maximum measured concentration of the analyte) | up to 20 days
Part A: AUC0-tz (area under the concentration-time curve of the analyte over the time interval from 0 to the last quantifiable time point) | up to 20 days
Part B: Cmax | up to 6 days
Part B: AUC0-tz | up to 6 days

CONTACTS AND LOCATIONS:
Locations (1):
- ICON-Groningen-62040, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com